CLINICAL TRIAL: NCT05082740
Title: Recalculating Breast Cancer Risk and Exploring the Experience of Receiving Updated Breast Cancer Risk Estimates in Women With a Family History of Breast Cancer
Brief Title: FH-Risk 2.0: Updating Breast Cancer Risk Estimates
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Victoria Woof, Miss, University of Manchester
Other Study IDs: FH-Risk 2.0 Research Protocol
Record Dates: First submitted 2021-09-24; First posted 2021-10-19 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Risk

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with a family history of breast cancer: This women are register to the Family History Risk and Prevention clinic and have taken part in the original FH-Risk study. These women will be given the opportunity to learn of their revised breast cancer risk estimate.
  Interventions: Other: Notification of a revised breast cancer risk estimate

INTERVENTIONS:
Other: Notification of a revised breast cancer risk estimate — These women will be given the opportunity to learn of their revised breast cancer risk estimate which has been re-calculated with the inclusion of new strong independent risk factors. These women will be offered a clinical consultation to discuss their risk and will a subset will be asked to take part in a qualitative interview about their experiences.

SUMMARY:
In the UK women with a strong family history of breast cancer are eligible for breast cancer risk estimation via Family History Risk and Prevention Clinics (FHRPCs). Here breast cancer risk is calculated using popular risk prediction models like the Tyrer-Cuzick, CanRisk or Gail models. These models combine breast cancer risk factors to calculate a risk estimate for women. Risk factors include, family history, hormonal and reproductive factors, and risk factors related to health behaviours, for example, smoking, exercise and alcohol intake.

Recently, risk estimation for breast cancer has become more accurate with the inclusion of mammographic density and Single Nucleotide Polymorphisms (SNPs) into popular risk prediction models. The addition of these new risk factors could alter the risk estimates that women in FHRPCs have been provided. How much these new risk factors alter a previously given risk estimate is unknown. It is also unknown how women will react to a revised risk estimate, especially if it changes their previous estimate and their access to preventive management options.

This research aims to explore this gap in the literature.

DETAILED DESCRIPTION:
Estimation of breast cancer risk is important since it enables selection of a high and moderate risk population who benefit from more frequent breast screening and the introduction of targeted measures to reduce risk such as lifestyle change, chemoprevention and risk reducing surgery. Traditionally, risk is estimated by combining information concerning family history and non-familial factors, such as age of menarche and first pregnancy. Subsequent management is related to the degree of risk (high, moderate or average) according to NICE guidelines. Members of the research team and others have added mammographic density (MD) and breast cancer risk associated single nucleotide polymorphisms (SNPs) to risk models which improves the accuracy of risk estimation but which may change the original given risk and risk management given before the updated models became available.

The objective of this body of work is to quantify change in risk and risk management when MD and SNPs are incorporated into two standard models (Tyrer-Cuzick v8 & BOADACEA V). A second objective of the study is to determine the psychological effects of change of risk and management.

This work will use participant data from the Family History Risk (FH-Risk) study to recalculate risk. The FH-Risk study population consists of 954 women referred to the Family History Risk and Prevention Clinic (FHRPC) between 2000 and 2012 who gave informed consent for DNA testing and estimation of MD as part of the FH-Risk study which recruited between 2010 and 2012. Change in risk and management will be calculated by comparing given risk at the time of clinic entry compared with re-estimated risk when MD and SNPs are added to the risk models according to NICE guidelines. Risk will be estimated retrospectively at the time of entry to the clinic and the time of latest follow up.

A sample of those who took part in the FH-Risk study who are still in the FHRPC for follow-up or discharged (approx.954) will be given the opportunity to discuss their updated risk.

Following the risk update consultation a sample of women will be asked whether they would like to take part in an interview to assess the psychological effects of the change, as well as their views and perceptions of the change. These interviews will inform the development of information materials for communicating recalculated risk. These materials will be appraised via 'think aloud' interviews with women from the FH-Risk study who have received their recalculated risk.

The results of this work are likely to inform the next iteration of NICE management guidelines for Family History Clinics, as well as inform the creation of patient facing information materials to aid patient - healthcare professional communication. The findings will also be used to develop a questionnaire to be given to women who previously took part in the FH-Risk study to assess the psychological impact of changed risk in a definitive study.

This body of work is split into 3 studies:

Study 1 - risk recalculation

Risk recalculation will be performed for all women who took part in the original FH-Risk study, with all women (still under follow up at the FHRPC or discharged) given the opportunity to attend a consultation to discuss their revised breast cancer risk estimate.

Study 2 - women's experiences of receiving a revised breast cancer risk estimate.

One to one semi-structured interviews will be conducting with women from study 1 to explore their experiences of receiving a revised breast cancer risk estimate. Breast cancer risk appraisals, the trustworthiness of the estimate, women's emotional responses will all be considered in these interviews. Information and communication needs will also be explored.

Study 3 - a questionnaire study assessing for whether women's subjective risk appraisals are inline with the revised risk estimate provided.

A questionnaire will be distributed to women in the study and they will be asked about their subjective risk appraisals, their thoughts on whether risk has changed, their satisfaction with the risk communicated and their cancer worry.

ELIGIBILITY:
Inclusion Criteria:

* previously given informed consent to participate in the original FH-Risk study,
* have an up to date clear mammogram,
* aged between 25 and 60,
* have not developed breast cancer and,
* have the capacity to consent.

Exclusion Criteria:

* women who have received a diagnosis of breast cancer,
* women who have not had a clear mammogram,
* women who took part in the original FH-Risk study but did not consent for their data to be used in future research and,
* women who lack the capacity to consent.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must identify as a woman and be born female
Study Population: Women in study will have taken part in the original FH-Risk study and who are still under follow up at the family history clinic or who have been discharged. These women will have had no history of breast cancer themselves. Women will be between the ages of 25 and 60.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
To explore how much new risk models change breast cancer risk estimates | 1 - 2 years
  How do new risk models which include mammographic density, SNPs and mutation testing change breast cancer risk estimates in women who are still registered at the family history clinic. Scatterplots and correlation coefficients will be used to examine the relationships between models and Bland-Altman plots used to show the agreement between the models.
To compare breast cancer risk models | 1 - 2 years
  Comparing the risk estimations given by the Tyrer-Cuzick and CanRisk models. Scatterplots and correlation coefficients will be used to examine the relationships between models and Bland-Altman plots used to show the agreement between the models.
To explore women's risk appraises and experiences of receiving a revised breast cancer risk estimate | Through to study completion, 2.5 years
  How do women react to receiving a revised breast cancer risk estimate, especially if their risk has changed. What are their risk perceptions following a revised estimate. This will assessed through qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Evans, Principal Investigator — Manchester University NHS Foundation Trust; Anthony Howell, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data from the study will be shared with other researchers on request. Data will included, an anonymised data set of women's breast cancer risk and anonymised interview transcripts. Women in the study will not be identifiable to other researchers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT05082740/Prot_SAP_000.pdf